CLINICAL TRIAL: NCT00865540
Title: Effect of Anti-inflammatory Topical Prednisolone Acetate 1%, Nepafenac of 0.1% and Ketorolac Tromethamine 0.4% in Intra-operative Mydriasis in Facetectomies
Brief Title: Effect of Anti-inflammatory Topical Prednisolone, Nepafenac and Ketorolac in Intra-operative Mydriasis in Facetectomies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Oftamologica Zona Sul (Other)
Responsible Party: Alexandre Paashaus da Costa Pinto, Clínica Oftalmológica Zona Sul
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OMB NO:0925-0586
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2009-03

CONDITIONS: Cataract
Keywords: cataract; pupillary dilation; anti-inflammatory; therapeutic use
MeSH Terms: conditions — Cataract; Mydriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- prednisolone acetate 1% (Experimental): one drop every 8h two days before surgery
  Interventions: Drug: prednisolone acetate 1%
- ketorolac tromethamine 0.4% (Experimental): one drop every 8h two days before surgery
  Interventions: Drug: ketorolac tromethamine 0.4%
- nepafenac 0.1% (Experimental): one drop every 8h two days before surgery
  Interventions: Drug: nepafenac 0.1%
- placebo (Placebo Comparator): one drop every 8h two days before surgery
  Interventions: Drug: methylcellulose 0.5%

INTERVENTIONS:
Drug: prednisolone acetate 1% — 1 drop every 8h two days before surgery
  Arms: prednisolone acetate 1%
Drug: ketorolac tromethamine 0.4% — 1 drop every 8h two days before surgery
  Arms: ketorolac tromethamine 0.4%
Drug: nepafenac 0.1% — 1 drop every 8h two days before surgery
  Arms: nepafenac 0.1%
Drug: methylcellulose 0.5% — 1 drop every 8h two days before surgery
  Arms: placebo

SUMMARY:
The main objective of this study is to compare the effect of preoperative use of anti-inflammatory topical prednisolone acetate 1%, nepafenac 0.1% and ketorolac tromethamine 0.4% of, plus a placebo, in maintaining the intra-operative mydriasis in extraction.

DETAILED DESCRIPTION:
Will be conducted with a randomized clinical trial volunteers with indication of extraction in Recife, Brazil. The surgical technique is employed phacoemulsification with implantation of intraocular lens. Digital photos are taken of the eye at the beginning and end of surgery and with them will be digitally determined the relationship between the corneal area and pupillary area. Each volunteer will be drawn to one of four groups of study (group 1, prednisolone acetate 1%, group 2, of ketorolac tromethamine 0.4%, 0.1% nepafenac group 3 and group 4, placebo). For the volunteers randomly selected for each group will be prescribed medication in its presentation as eye drops (Prednisolone acetate 1%, Pred Fort ®, Allergan ®; of ketorolac tromethamine 0.4%, incite l ®, Allergan ®; Nepafenac 0.1%, Nevanac ® Alcon ® and 0.5% methylcellulose, Fresh Tears ®, Allergan ®), 01 drop every 8 hours for 48 hours before surgery. For all volunteers will also be prescribed gatifloxacin (Zymar ®), 01 drop every 8 hours starting 48 hours before surgery. Was scheduled a minimum sample of 60 volunteers (15 per group).

ELIGIBILITY:
Inclusion Criteria:

* Carriers of senile cataract (> 50 years of age) with indication for cataract extraction with implantation of intraocular lens, with local anesthesia

Exclusion Criteria:

* Diabetic
* Using systemic anti-hormonal and non-hormonal
* Using topical ocular medication (including anti-glaucomatous)
* Individuals with congenital ocular abnormalities and cases in which there is intra-operative complications (hernia or trauma in the iris, posterior capsule rupture or zônula and prolonged phacoemulsification time of ≥ 1 minute).
* Volunteers with incipient nuclear cataract (density 1) or advanced (density 4) by the LOCS II classification (density of nuclear cataract ranked 1 to 4 (Chalk et al, 1989)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
pupil size | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre P Costa, Pinto, Principal Investigator — Clínica Oftalmológica Zona Sul
Locations (1):
- Clínica Oftalmológica Zona Sul, Recife, Pernambuco, Brazil